CLINICAL TRIAL: NCT03357588
Title: Evaluation of an Intensified Treatment Monitoring Strategy to Prevent Accumulation and Spread of HIV-1 Drug Resistance in Low- and Middle-income Countries (ITREMA).
Brief Title: The Intensified Treatment Monitoring Strategy to Prevent Accumulation of Drug Resistance (ITREMA) Trial
Acronym: ITREMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Ndlovu Care Group (Unknown); Wits Reproductive Health and HIV Institute (Other)
Responsible Party: Principal Investigator, Dr. Annemarie Wensing, Clinical Virologist, Head of Medical Microbiology Residency Program, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69/2015
Record Dates: First submitted 2017-09-28; First posted 2017-11-30 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Standard of Care monitoring
  Interventions: Other: Standard of care monitoring
- Intervention (Experimental): Intensified monitoring
  Interventions: Other: Intensified monitoring

INTERVENTIONS:
Other: Intensified monitoring — Intensified virological monitoring during first-line ART with viral load monitoring at month 6 of ART and 3-monthly thereafter, followed-up consecutively by point-of-care qualitative drug level testing and drug resistance testing in case of a viral load >1000 copies/mL, during first-line antiretroviral treatment (ART) for HIV-1 infection as prescribed by South African national guidelines.
  Arms: Intervention
Other: Standard of care monitoring — Standard-of-care virological monitoring during first-line ART as described by WHO and South African National Department of Health ART guidelines, consisting of viral load monitoring at month 6 and 12 of ART and annually thereafter, followed-up by a repeat measurement within 3 months after a viral load >1000 copies/mL, during first-line antiretroviral treatment (ART) for HIV-1 infection as prescribed by South African national guidelines.
  Arms: Control

SUMMARY:
The ITREMA trial is an open-label randomized controlled trial (RCT) in which HIV-1 infected patients initiating first-line ART and already on first-line ART will be enrolled. Enrollment will continue until 600 patients have been randomized. Patients initiating ART will be randomized after six months of ART and patients already on ART will be randomized at 6 months after the last viral load measurement. Patients in both arms will receive study visits every three months for a total follow-up duration of 18 months after randomization to either of two study arms. The control arm will receive standard of care HIV-1 treatment monitoring during first-line ART in accordance with South African National Department of Health (NDoH) guidelines. The intervention arm will receive intensified treatment monitoring during first-line ART according to the treatment monitoring strategy under investigation.

DETAILED DESCRIPTION:
This study will enroll adult HIV-1 infected patients who are about to initiate or have already initiated first-line ART. Patient enrollment and randomization will be performed at two different time points. Timing and criteria for enrollment and randomization are as follows:

1. ART naïve patients: Patients are eligible for enrollment initiation of treatment with first-line ART. Randomization is performed after availability of the first routine viral load measurement, performed at month 6 of treatment.
2. Patients on ART: Patients are eligible for enrollment after ≥ 1 year of virologically suppressive first-line ART and only if a last viral load with a result <1000 copies/mL was performed within the last 6 months. Randomization is performed 6 months after the last viral load (VL) result.

A total number of 600 patients will be randomized into two trial arms. The trial will be conducted on-site at one of the clinical facilities of Ndlovu Care Group (http://www.ndlovucaregroup.co.za/), one of the partners in the project. This facility, Ndlovu Medical Centre, is situated in the town of Elandsdoorn, Limpopo, South Africa, and provides medical service to local South African patients who are unable to pay medical insurance. The Ndlovu Care Group distributes antiretroviral medication in the framework of the South African Department of Health antiretroviral treatment programme. This clinic is currently providing ART to >3600 patients. Patients on ART return to the clinic monthly for collection of medication, pill count and adherence counselling, which allows intensification of monitoring without substantial change of the infrastructure or frequency of visits.

After randomisation, patients in both study arms will return for study follow-up visits on a three-monthly basis, at month 9, 12, 15, 18, 21 and 24 after start of ART or after the last VL measurement. In addition, patients will be called back for additional study visits (max. 2) in case of a detected viral load >1000 copies/ml during any of these visits. All visits in both arms, including aforementioned additional call back visits will coincide with standard of care medication collection visits to the clinic. In case of a switch to second-line therapy, patients in both arms will continue three-monthly follow-up visits in an observational manner, and guidelines for monitoring of second-line therapy are followed.

Control arm:

300 patients randomly assigned to this arm will be monitored in full concordance with current South African NDoH guidelines in use at the study site. Viral load measurements will be performed at month 12 and 24 after start of ART (for newly initiated patients) or at month 12 and 24 after the last viral load measurement (patients already on ART). If a viral load >1000 copies/ml is detected, the patient is called back for counseling for therapy adherence and repeat viral load measurement, 2 months after the initial viral load measurement. If the repeat viral load measurement is >1000 copies/ml after adherence counseling, this is taken to be indicative of therapy failure due to development of drug resistance and a switch to second line therapy is made, together with intensified adherence counseling, without verifying the cause of virological failure by performing drug level testing or drug resistance testing. If viral load drops to <1000 copies/ml after adherence counseling, the first line treatment is maintained.

Intervention arm:

300 patients randomly assigned to this arm will be monitored using the investigational intensified monitoring strategy. This strategy consists of 3-monthly viral load monitoring at month 9, 12, 15, 18, 21 and 24 (after start of ART in initiating patients or after the last viral load measurement in patients on ART). If a viral load measurement > 1000 copies/mL is detected, the patient will be called back for a follow-up study visit at the next monthly medication collection visit (4 weeks after detection of elevated viral load). Upon arrival drug level testing is performed, the viral load measurement is repeated, and a dried blood spot prepared and stored at room temperature. Procedures following this depend on the result of drug level testing:

* If drug levels are detected by drug level testing, the result of the viral load measurement is awaited. If the repeat viral load is >1000 copies/ml, the dried blood spot is shipped directly by courier to the World Health Organization (WHO) reference laboratory for drug resistance testing. The reference laboratory will provide feedback by means of a digital resistance report to the coordinating research physician. The patient will be called back for a second follow-up study visit at the next monthly medication visit (8 weeks after detection of elevated viral load), either for prescription of second-line therapy or continuation of first-line therapy, guided by the result of resistance testing.
* If drug level monitoring at the first follow-up visit indicates that drug levels are not detected, intensified counseling is performed at the same visit and first-line therapy will be maintained, regardless of the result of the repeat viral load measurement. The patient will not be called back and the next viral load will be performed at the next scheduled three-monthly time point. However, if the viral load result at this visit is again >1000 copies/ml, drug resistance testing will be performed regardless of the outcome of drug level testing.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected male or female patients
* For ART Naïve patients: Eligible for and intending to initiate ART at the clinical site
* For patients on ART: On ART ≥1 year. Last VL <6 months ago and <1000 copies/mL
* ≥18 years of age
* Able to understand and willing to give informed consent

Exclusion Criteria:

* Any serious unstable medical condition at study baseline
* Any criteria that in the opinion of the investigator indicate that the patient is unable to participate in the full study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
Drug resistance | week 48
  Prevalence of drug resistance in patients with therapy failure in each arm
Drug resistance | week 96
  Prevalence of drug resistance in patients with therapy failure in each arm
Unnecessary treatment switches | week 48
  Number of virological failure cases without drug resistance in the intervention arm (averted unnecessary treatment switches) versus in the control arm (unnecessary treatment switches)
Unnecessary treatment switches | week 96
  Number of virological failure cases without drug resistance in the intervention arm (averted unnecessary treatment switches) versus in the control arm (unnecessary treatment switches)

SECONDARY OUTCOMES:
Time on failing regimen | week 96
  Time during which viremia > 1000 copies/mL is maintained after the first instance of a viral load >1000 copies/ml
Loss of second line therapeutic options over time | week 96
  The loss of second line therapeutic options over time due to accumulation of resistance mutations in the presence of a failing regimen.
Influence of genotypic resistance testing | week 96
  Influence of genotypic resistance testing on the choice for a second line regimen by comparing chosen regimens in the intervention and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Annemarie MJ Wensing, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- Ndlovu Medical Centre, Elandsdoorn, Limpopo, South Africa

REFERENCES:
- [Derived] Gumede SB, Wensing AMJ, Lalla-Edward ST, de Wit JBF, Francois Venter WD, Tempelman HA, Hermans LE. Predictors of Treatment Adherence and Virological Failure Among People Living with HIV Receiving Antiretroviral Therapy in a South African Rural Community: A Sub-study of the ITREMA Randomised Clinical Trial. AIDS Behav. 2023 Dec;27(12):3863-3885. doi: 10.1007/s10461-023-04103-2. Epub 2023 Jun 29. PMID 37382825
- [Derived] Hermans LE, Nijhuis M, Tempelman HA, Houts T, Schuurman R, Burger DM, Wensing AMJ, ter Heine R. Point-of-Care Detection of Nonadherence to Antiretroviral Treatment for HIV-1 in Resource-Limited Settings Using Drug Level Testing for Efavirenz, Lopinavir, and Dolutegravir: A Validation and Pharmacokinetic Simulation Study. J Acquir Immune Defic Syndr. 2021 Aug 1;87(4):1072-1078. doi: 10.1097/QAI.0000000000002681. PMID 34153013